CLINICAL TRIAL: NCT06116968
Title: An Open-Label Study of Aficamten for Chinese Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: An Open-Label Study of Aficamten for Chinese Patients With Symptomatic oHCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX01003; CTR20233249 (Registry Identifier: China Center for Drug Evaluation(CDE))
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aficamten (Experimental): Patients in this arm take daily dose of Aficamten. Each patient will start at the lowest dose (5 mg) in the pre-specified dose range and undergo dose titration up to a maximum of 20 mg.
  Interventions: Drug: Aficamten

INTERVENTIONS:
Drug: Aficamten — 5-20mg
  Other Names: CK-3773274

SUMMARY:
This is an open-label extension study of China cohort in the phase 3 study (CY 6031) of aficamten for the treatment of obstructive HCM (oHCM) to collect long-term safety and tolerability data, including assessments of cardiac function and steady-state Pharmacokinetics (PK) during chronic dosing with aficamten.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of a Cytokinetics trial investigating CK-3773274
2. LVEF ≥55% at the Screening Visit

Exclusion Criteria:

1. Has participated in another investigational device or drug study or received an investigational device or drug <1 month (or 5 half-lives for drugs, whichever is longer) prior to screening. Other investigational procedures while participating in this study are not permitted.
2. Since completion of a previous study of aficamten has:Developed new-onset paroxysmal or permanent atrial fibrillation (AF) requiring rhythm restoring treatment (e.g., direct-current cardioversion, ablation procedure, or antiarrhythmic therapy) <30 days prior to screening. Patient may rescreen for JX01003 after 30 days if heart rate (HR) <100 bpm and/or rhythm is stable >30 days.
3. Undergone septal reduction therapy (surgical myectomy or transcatheter alcohol ablation).
4. Had a confirmed LVEF <40% with an associated dose interruption during participation in a prior study with aficamten.
5. History of appropriate implantable cardioverter defibrillator (ICD) shock within 30 days prior to screening.
6. Has received treatment with mavacamten.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Patient incidence of reported adverse events (AEs) | Baseline to End of study, up to 2 years
Patient incidence of reported serious adverse events (SAEs ) | Baseline to End of study, up to 2 years
Patient incidence of LVEF<50% & LVEF <40% | Baseline to End of study, up to 2 years

SECONDARY OUTCOMES:
Peak LVOT-G at rest and with Valsalva provocation | Change from baseline values to week 48 at 12-week intervals;
Proportion of patients with resting LVOT-G <50 mmHg | Change from baseline values to week 48 at 12-week intervals;
Proportion of patients with resting LVOT-G <30 mmHg | Change from baseline values to week 48 at 12-week intervals;
Proportion of patients with post-Valsalva LVOT-G <50 mmHg | Change from baseline values to week 48 at 12-week intervals;
Proportion of patients with post-Valsalva LVOT-G <30 mmHg | Change from baseline values to week 48 at 12-week intervals;
Proportion of patients with LVEF ≥50%, resting LVOT-G <30 mmHg, and post-Valsalva LVOT-G <50 mmHg | Change from baseline values to week 48 at 12-week intervals;
First resting LVOT-G <50 mmHg | Time to the following event through last follow-up, up to 2 years.
First resting LVOT-G <30 mmHg | Time to the following event through last follow-up, up to 2 years.
First post-Valsalva LVOT-G <50 mmHg | Time to the following event through last follow-up, up to 2 years.
First post-Valsalva LVOT-G <30 mmHg | Time to the following event through last follow-up, up to 2 years.
First LVEF ≥50%, resting LVOT-G <30 mmHg, and post-Valsalva LVOT-G <50 mmHg | Time to the following event through last follow-up, up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhui Zhang, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (12):
- China (12):
  - Beijing Anzhen Hospital, Beijing
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing
  - Fuwai Hospital, CAMS & PUMC, Beijing
  - Peking University Third Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - Nanfang Hospital, Guangzhou
  - The Second Affiliated Hospital of Nanchang University, Jiangxi
  - The First Hospital of Jilin University, Jilin
  - Shengjing Hospital of China Medical University, Shenyang
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No